CLINICAL TRIAL: NCT01567553
Title: Early Neuroinflammatory Changes as a Prognostic Marker in Clinically Isolated Syndromes Patients.
Brief Title: The Inflammatory Process and the Medical Imaging in Patients With an Inflammatory Disease of the Central Nervous System.
Acronym: USPIO-CIS
Status: Terminated | Type: Observational
Why Stopped: terminated ( Halted prematurely,expiration of investigationnal product)
Sponsor: Rennes University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007-005363-10
Record Dates: First submitted 2012-02-24; First posted 2012-03-30 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis (MS); Inflammatory Disease
Keywords: inflammatory disease of the central nervous system; early clinical deficit; multiple sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Only unenhanced MR scanning will be performed in a control group of normal, age-matched subjects and after acceptance of the protocol by an independent ethical committee for the implication of a normal population in such an MRI research project.
  Interventions: Other: USPIO MRI - Gadolinium MRI
- Experimental group: CIS at presentation (clinically isolated syndromes) will be recruited with MRI evidence of at least two asymptomatic brain MRI lesions. The group will compromise 50 CIS patients. These CIS patients will be included within three months after first clinical presentation.
  Interventions: Other: USPIO MRI - Gadolinium MRI

INTERVENTIONS:
Other: USPIO MRI - Gadolinium MRI — USPIO MRI scanning will be performed at :
  * baseline, month 3, month 6, month 9 and month 12 for patients recruited prior to the 1st of May 2010.
  * baseline, month3, month 6 and month 9 for patients recruited between the 1st of May 2010 and the 31st of July 2010,
  * baseline, month 3 and month 6 for patients recruited between the 1st of August 2010 and the 31st of October 2010,
  * baseline and month 3 for patients recruited between the 1st of November 2010 and the 31st of January 2011,
  * baseline for patients recruited between the 1st of February 2011 and the 30rd of April 2011.
  Gadolinium MRI scanning will be performed at baseline, month 3, month 6, month 9, month 12, month 18, month 24 and month 36.

SUMMARY:
While significant progress has been made on medical imagery in recent years in the individualization of different lesions in the nervous system for demyelination, axonal loss, atrophy, little progress has been made in the specific recognition the inflammatory process. Yet this point is essential since the currently available treatments have a partial impact mainly on the inflammatory component and that many uncertainties remain about the links between inflammation and tissue destruction affecting myelin and axons. The recent discovery of a macrophage cell marker in the CNS, more specific (USPIO) of inflammation gives us the opportunity to answer important questions which one can sense that this could have a significant impact on therapeutic drug monitoring of these patients. This study will involve 50 patients recruited in five French centers (Marseille, Paris, Reims, Rennes, Toulouse) from the earliest manifestations of the disease with clinical and MRI scheduled for the first 3 years of their disease.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system affecting 60.000 persons in France and characterized by widespread inflammation, focal demyelination, and a variable degree of axonal loss. In recent years the concept of MS as an inflammatory neurodegenerative disease has been corroborated by neuropathologic and in vivo MR imaging studies. A number of MR studies show that the principal pathological substrate of permanent disability is axonal loss as detected in MR studies as global atrophy, but also regionally in the white or grey matter, and that atrophy already occurs at early stages of the disease. Though MR imaging is a powerful tool for MS in terms of diagnosis, description of the natural history of the disease and treatment monitoring, the major drawback of MRI in MS is the lack of specificity of the MR findings. Furthermore, with the advent of disease modifying drugs, there is a need for robust and specific MR markers to identify e.g. clinically isolated syndrome (CIS) patients at presentation at high risk to develop MS or a more severe disease course. An increasing body of MRI evidence corroborates that CIS show early and dynamic changes detected by MR imaging, such as global or regional brain atrophy, as a sign of progressive axonal loss, but atrophy is already a late stage sign of the disease, when tissue is lost. Considerable efforts are spent today to identify early and prognostic MR markers for high risk CIS patients.

In the current project we endeavour to study CIS patients with inflammatory disease of the central nervous system or early clinical deficit by using cell labelling MR imaging with ultra small superparamagnetic iron oxide particles (USPIO), which specifically label blood-borne macrophages, a key cell population in MS. We hypothesise that number/volume of USPIO (SH U 555 C) enhancement during the first year is a predictive marker for high risk CIS patients at presentation. This hypothesis is in line with recent findings in the animal model of MS, EAE. Secondary measures of this study will include comparison of the USPIO (SH U 555 C) findings with other highly sensitive, but non-specific MR parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Patients with a first episode suggestive of MS (monofocal or multifocal)
* Presence of a first neurologic event suggestive of MS that lasted for at least 24 hours
* Patients with a spatial dissemination criteria according to the Mc Donald diagnostic criteria
* With an Expanded Disability Status Scale (EDSS) score at baseline between 0 and 5
* USPIO (SH U 555 C) injection has to be performed within 3 months after start of clinical event
* Patients have to be in-patients for a minimum of 24 hours after the first USPIO (SH U 555 C) injection
* Patients with positive or negative USPIO-MRI during screening are included
* Patients must be compliant with study protocol
* Patients must have given their written consent to participate in this study

Exclusion Criteria:

* Any CIS patients having received steroid treatment before acquisition of the baseline USPIO MR scan
* Patients in whom any disease other than MS could explain their signs and symptoms,
* Patients with complete transverse myelitis or bilateral optic neuritis will be excluded,
* Patients who had received prior immunosuppressive or immunomodulatory treatment will be excluded.
* Patients who had received corticoids 30 days before USPIO-RMI
* Patients which cannot be in-patients for a minimum of 24 hours after the first USPIO (SH U 555 C) injection
* Female patients without efficient contraception (oral or others) Pregnant or lactating patients
* Patients with a known allergy to iron particles and/or dextrans
* Patients having received in the past 5 months iron oxide particles preceding the MRI examination
* Patients with a past history of bronchial asthma or any other allergic disorder
* Patients with a past history for a lower threshold of seizures
* Any patient presenting with a known contra-indication for MR scanning
* Non-compliant or uncooperative patients with regard to study protocol
* Patients not having given their written consent to participate in this study
* Any patient with an accompanying systemic disease, renal disease, cardiac disease or mental disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: CIS at presentation (clinically isolated syndromes) will be recruited with MRI evidence of at least two asymptomatic brain MRI lesions. The group will compromise 50 CIS patients. These CIS patients will be included within three months after first clinical presentation.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
▪ Change in USPIO enhancing MS lesion | Change from baseline in USPIO enhancing MS lesion at 12 months after the first event of the disease
  USPIO enhancing MS lesion at baseline and during 12 month after the first event of the disease as a predictor for a higher risk to develop a second clinical event (time to second clinical event) in CIS patients (evidence of USPIO enhancement: yes/no; and number of USPIO lesions).

SECONDARY OUTCOMES:
Comparison of primary outcome measures with clinical outcomes and role of USPIO | at 12 months after the first event of the disease
  ▪ Comparison of primary outcome measures with clinical outcomes (EDSS and conversion to MS) - and role of USPIO (SH U 555 C) as a potential biomarker to predict these two clinical outcomes
Relationship of USPIO (SH U 555 C) enhancing MRI lesions with other MR parameters | at 12 months after the first event of the disease
  ▪ Relationship of USPIO (SH U 555 C) enhancing MRI lesions with other MR parameters (Differently weighted MR-lesions : T2, T1, FLAIR ; MR diffusion measures, MTR ; MR atrophy measures (global and regional atrophy))
Change in USPIO and/or Gadolinium enhancing MS lesions (primary outcome measure) | Change from baseline in USPIO and/or Gadolinium enhancing MS lesions at 3 years after the first event of the disease
  ▪ USPIO and/or Gadolinium enhancing MS lesions as a predictor for a higher risk to develop a second clinical event (time to second clinical event) in CIS patients (evidence of USPIO or Gd enhancement: yes/no; and number of USPIO and/or Gd lesions)at 3 years after the first event of the disease

CONTACTS AND LOCATIONS:
Overall Officials: EDAN Gilles, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - La Timone University Hospital (APHM), Marseille
  - La Pitie-Salpaetriere Hospital (APHP), Paris
  - Maison Blanche Hospital, Reims
  - Rennes University Hospital, Rennes
  - Purpan Hospital, Toulouse

REFERENCES:
- [Result] Crimi A, Commowick O, Maarouf A, Ferre JC, Bannier E, Tourbah A, Berry I, Ranjeva JP, Edan G, Barillot C. Predictive value of imaging markers at multiple sclerosis disease onset based on gadolinium- and USPIO-enhanced MRI and machine learning. PLoS One. 2014 Apr 1;9(4):e93024. doi: 10.1371/journal.pone.0093024. eCollection 2014. PMID 24691080